CLINICAL TRIAL: NCT02653885
Title: Haematologic Predictors and Clinical Outcome in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, MD, Ankara University
Other Study IDs: YIH
Record Dates: First submitted 2016-01-11; First posted 2016-01-12 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cardiac Disease
Keywords: cardiac surgery; open heart surgery; hemogram
MeSH Terms: conditions — Heart Diseases | interventions — Erythrocyte Indices; Mean Platelet Volume; Platelet Count

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Red red cell distribution width — Results from hemogram
  Other Names: Mean platelet volume; Platelet/lymphocyte ratio; Neutrophil/lymphocyte ratio

SUMMARY:
The outcome predictors for cardiac surgery has been popular for many researchers and clinicians. Determining risk factors before surgery reduce morbidity and mortality after surgery. Some routine blood results have been used as predictors for cardiac surgery but none of the researches studied red cell distribution width, mean platelet volume, platelet/lymphocyte ratio and neutrophil/lymphocyte ratio. This study focused on these parameters and to see whether these parameters can be predictors for cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective, on-pump cardiac surgery

Exclusion Criteria:

* emergent cases
* pediatric cases
* congenital surgery
* heart transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac patients needed cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
incidence of combined adverse effects | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, MD, Study Chair — Ankara University